CLINICAL TRIAL: NCT06539819
Title: Electrical Posterior Box Isolation and Rotor Modulation Ablation Versus Electrical Posterior Box Isolation Alone for the Treatment of Persistent Atrial Fibrillation
Brief Title: Rotor Modulation Ablation for the Treatment of Persistent Atrial Fibrillation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-KY-048
Record Dates: First submitted 2024-06-04; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-06

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical Posterior Box Isolation and Rotor Modulation Ablation group (R&B group) (Experimental): The subject's surgical procedure is electrical posterior box isolation plus rotor modulation ablation.
  Interventions: Procedure: Electrical Posterior Box Isolation and Rotor Modulation Ablation group (R&B group)
- Electrical Posterior Box Isolation group (BO group) (Active Comparator): The subject's surgical procedure is electrical posterior box isolation.
  Interventions: Procedure: Electrical Posterior Box Isolation group (BO group)

INTERVENTIONS:
Procedure: Electrical Posterior Box Isolation and Rotor Modulation Ablation group (R&B group) — the intervention is conducting electrical posterior box isolation plus rotor modulation ablation
  Arms: Electrical Posterior Box Isolation and Rotor Modulation Ablation group (R&B group)
Procedure: Electrical Posterior Box Isolation group (BO group) — the intervention is conducting electrical posterior box isolation alone
  Arms: Electrical Posterior Box Isolation group (BO group)

SUMMARY:
For Persistent atrial fibrillation (PeAF), the therapeutic effect of catheter ablation needs to be further improved. 3.Circumferential pulmonary vein isolation (CPVI) is the cornerstone of catheter ablation of AF, and additional ablation methods such as linear ablation or fragmentation potential ablation plus CPVI have been demonstrated to improve the treatment effect of PeAF, but there is still a large gap with the ideal ablation treatment effect.Recent studies have shown that the "rotor" is an important mechanism for the maintenance of PeAF, and related studies have shown that rotor modulation ablation may further improve the success rate of catheter ablation for PeAF. However, on the one hand, there is a lack of effective mapping catheter tool for rotor mapping, and on the other hand, the reproducibility of some related studies still needs to be further confirmed, and further clinical studies are needed to explore whether rotor modulation ablation can improve the success rate of catheter ablation for PeAF. The EnSite™ LiveView dynamic mapping system, combined with the HD Grid mapping catheter, provides a effective mapping tool for clinical surgeons. In the early clinical practice, we successfully completed the rotor mapping ablation using the mapping system, and there was no complication during the operation, which was safe and reliable, and achieved good intraoperative and postoperative results. We intend to conduct this clinical study to explore whether rotor ablation combined with BOX ablation can further improve the efficacy of PeAF compared with BOX ablation alone, and provide guidance for catheter ablation treatment of PeAF. This is a single-center, randomized, parallel-controlled, single-blind clinical trial, and we plan to enroll 360 subjects randomized into Electrical Posterior Box Isolation and Rotor Modulation Ablation group (R&B group) and Electrical Posterior Box Isolation group (BO group), The corresponding surgery was performed according to the group, and the postoperative follow-up was 12 months, and the main observation endpoint was the remission rate of atrial fibrillation one year after surgery.

DETAILED DESCRIPTION:
1. Atrial fibrillation (AF) is a common arrhythmia, and its incidence increases with age. In addition, AF is extremely harmful, and studies have found that AF significantly increases mortality, affects cardiac function, increases the risk of arterial embolism (e.g., stroke), and reduces quality of life. For rhythm control of AF, catheter ablation has been shown to be superior to medical therapy.
2. Persistent atrial fibrillation (PeAF) is one type of AF that lasts longer than 7 days and includes episodes that are terminated by cardioversion (medical or electrical cardioversion) after more than 7 days. For PeAF, the therapeutic effect of catheter ablation needs to be further improved.
3. Circumferential pulmonary vein isolation (CPVI) is the cornerstone of catheter ablation of AF, and additional ablation methods such as linear ablation or fragmentation potential ablation plus CPVI have been demonstrated to improve the treatment effect of PeAF, but there is still a large gap with the ideal ablation treatment effect. The reason of this dilemma is that the mechanism of occurrence and maintenance of AF is very complex, which has not yet been fully clarified.
4. Recent studies have shown that the "rotor" is an important mechanism for the maintenance of PeAF, and related studies have shown that rotor modulation ablation may further improve the success rate of catheter ablation for PeAF.
5. However, on the one hand, there is a lack of effective mapping catheter tool for rotor mapping, and on the other hand, the reproducibility of some related studies still needs to be further confirmed, and further clinical studies are needed to explore whether rotor modulation ablation can improve the success rate of catheter ablation for PeAF.
6. The EnSite™ LiveView dynamic mapping system, combined with the HD Grid mapping catheter, provides a effective mapping tool for clinical surgeons. The planar design of the HD Grid mapping catheter allows it to fit perfectly against the endocardium; The multi-directional perception function enables it to overcome the problem of bipolar blind spots. The EnSite™ LiveView dynamic mapping system can help the surgeon determine the process and time point of each potential activation by uploading the dynamic rhythm in real time, achieving better catheter stability compared to traditional mapping systems, eliminating the need for secondary mapping or saving of mapping points, and direct data interpretation when used with HD Grid catheters, which gives it a strong advantage over other mapping electrodes in the mapping rotor.
7. In the early clinical practice, we successfully completed the rotor mapping ablation using the mapping system, and there was no complication during the operation, which was safe and reliable, and achieved good intraoperative and postoperative results.
8. At present, for PeAF, our center generally uses BOX ablation, which is also one of the mainstream surgical methods for the treatment of PeAF in clinical practice. We intend to conduct this clinical study to explore whether rotor ablation combined with BOX ablation can further improve the efficacy of PeAF compared with BOX ablation alone, and provide guidance for catheter ablation treatment of PeAF.
9. This is a single-center, randomized, parallel-controlled, single-blind clinical trial, and we plan to enroll 360 subjects randomized into Electrical Posterior Box Isolation and Rotor Modulation Ablation group (R&B group) and Electrical Posterior Box Isolation group (BO group), The corresponding surgery was performed according to the group, and the postoperative follow-up was 12 months, and the main observation endpoint was the remission rate of atrial fibrillation one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinical Diagnosed of persistent atrial fibrillation； 2. Has an indication for radiofrequency ablation surgery and no contraindications to radiofrequency ablation (according to Current knowledge and management of atrial fibrillation: consensus of Chinese experts 2021)；3. Patients between the ages of 20 and 80 years, male or female；4. Left atrial systolic anteroposterior diameter (LAs)<55mm measured by thoracic ultrasound； 5. Patients who agree to undergo clinical trials and comply with the protocols, voluntarily sign the informed consent form.

Exclusion Criteria:

* 1. History of previous radiofrequency ablation of atrial fibrillation; 2. Left ventricular ejection fraction (LVEF) < 30% measured by thoracic ultrasound; 3. Cardiac surgery within the previous 180 days or expecting cardiac surgery within 180 days; 4. Coronary PTCA/stenting within the previous 90 days; 5. Patients with severe pulmonary, hepatic and renal insufficiency; 6. Diagnosed atrial myxoma; 7. Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment; 8. Women who are pregnant or who plan to become pregnant during the study; 9. Acute illness or active infection at time of index procedure; 10. Acute coronary syndrome within the previous 60 days; 10. History of blood clotting or bleeding abnormalities; 12. Contraindication to anticoagulation; 13. Life expectancy less than 1 year; 14. Uncontrolled heart failure; 15. Presence of an intramural thrombus, tumor, or other abnormality that precludes catheter introduction or positioning; 16. Cannot be removed from antiarrhythmic drugs for reasons other than atrial fibrillation; 17. Unwilling or unable to provide informed consent; 18. Uncontrolled alcoholics; 19. Patients with hypertrophic cardiomyopathy; 20. Patients with poorly controlled hypertension (blood pressure >140/90 mmHg despite antihypertensive therapy).

Ages: 21 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The rate of freedom from AF within one year after surgery | 1, 3, 6, 12 months after surgery
  The rate of freedom from AF within one year after surgery

SECONDARY OUTCOMES:
Incidence of other atrial arrhythmias within one year after surgery | 1, 3, 6, 12 months after surgery
  Incidence of other atrial arrhythmias within one year after surgery
Cardiac function | 12 months after surgery
  Cardiac function was valued by left ventricular ejection fraction measured by transthoracic echocardiography
Incidence of thrombosis-related events | 12 months after surgery
  Incidence of thrombosis-related events
Serious complications associated with ablation procedure | 12 months after surgery
  Serious complications associated with ablation procedure